CLINICAL TRIAL: NCT00443833
Title: Genetic Analysis of Thai Patients With Thyrotoxic Periodic Paralysis
Brief Title: Genetic Analysis of Thyrotoxic Periodic Paralysis
Status: Completed | Type: Observational
Sponsor: Ramathibodi Hospital (Other)
Other Study IDs: 11-46-21
Record Dates: First submitted 2007-03-05; First posted 2007-03-06 (Estimated); Last update posted 2007-03-06 (Estimated); Status verified 2007-03

CONDITIONS: Thyrotoxic Periodic Paralysis
Keywords: Thyrotoxicosis; genetic association study; periodic paralysis; whole genome scan
MeSH Terms: conditions — Thyrotoxicosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
Thyrotoxic periodic paralysis (TPP) is characterized by episodes of reversible hypokalemia and weakness in thyrotoxic patients. It is commonly found in males of Asian descent and is also seen in individuals having Native American or Hispanic ancestry. Therefore genetic etiology has been hypothesized. This study, we aim to find the susceptibility genes that associate with TPP. Both candidate genes approach and genome wide association study have been conducted.

DETAILED DESCRIPTION:
This study is a genetic association study. It included 50 cases of TPP patients and 80 cases of male, hyperthyroid patients who didn't have hypokalemia as a well characterized controls. After informed consent were obtained, genomic DNA from leukocyte were extracted. Pooled DNA were constructed and whole genome scan using 10K GeneChip microarray were genotyped on pooled genomic DNA.

ELIGIBILITY:
Inclusion Criteria:

TPP

* Hyperthyroid patients from any causes
* Evidence of hypokalemia (k<3.5 mg/dl)from intracellular shift (Urine K<15 mg/dl, TTKG<2)
* Episodic paralysis

Exclusion Criteria:

* Hypokalemia from GI or renal loss

Min Age: 15 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80
Dates: Start 2004-01; Study Completion 2005-12

CONTACTS AND LOCATIONS:
Overall Officials: Wallaya Jongjaroenprasert, MD, Principal Investigator — Endocrinology Unit, Ramathibodi Hospital, Mahidol University